CLINICAL TRIAL: NCT06963567
Title: Observational Registry to Determine the Predictors and Outcomes of Patients at Risk of and Diagnosed With Left Ventricular Thrombus
Brief Title: Left Ventricular Thrombus Registry
Acronym: LVT Registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 336025; G-002409 (Other Grant/Funding Number: Barts Charity)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Left Ventricular Thrombus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LV Thrombus (present): Patients with a diagnosis of LV thrombus in the setting of LV dysfunction (acute myocardial infarction, Ischaemic Cardiomyopathy (ICM), dilated cardiomyopathy (DCM)).
- LV Thrombus (at risk): Patients that do not have LV thrombus but are at risk for developing thrombus such as those with severe LV dysfunction, LV aneurysms, large territory infarcts will also be included.

SUMMARY:
Left Ventricular Thrombus (LVT) is a blood clot that can develop in a poorly functioning heart. In around 1 in 6 patients who have had a heart attack or diagnosed with heart failure tend to develop blood clots in their main heart chamber.

Having a blot clot in the main heart chamber can lead to serious complications such as stroke. Treatment for blood clots is blood thinning medications, which if taken for a prolonged period of time can result in bleeding which further complicates treatment. We hope to gather information to better understand the factors associated with blood clot formation and management in the lower left chamber of the heart. This understanding will hopefully enable us and others to improve management of this condition in the future and therefore help the wider population. As part of this study, bloods and scan results will be recorded and we will complete a short quality of life questionnaire. When participants come in for routine MRI scan, we may capture additional images for further research analysis.

A sample of blood no more than one tablespoon will be collected for research analysis at the same time as routine blood test. This will occur at baseline and at around 6 months. At 12 months we will repeat the quality of life questionnaire and collect final data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LV thrombus or;
* Patients at risk for developing LV thrombus (e.g severe LV dysfunction, LV aneurysm, MI.

Exclusion Criteria:

* Age < 18 years
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of LV thrombus in the setting of LV dysfunction (acute myocardial infarction, Ischaemic Cardiomyopathy (ICM), dilated cardiomyopathy (DCM)) will be screened. Patients that do not have LV thrombus but are at risk for developing thrombus such as those with severe LV dysfunction, LV aneurysms, large territory infarcts will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite Result | From baseline to final 12 month follow up (+/- 2 months)
  To measure the composite result of major bleeding (BARC >3), stroke and systemic embolisation, and all-cause mortality

SECONDARY OUTCOMES:
CMR prediction of thrombus | From baseline to 6 month follow up (+/- 3 months)
  To assess CMR based risk prediction model of recurrence of LV thrombus
Blood Test | From baseline to 6 month follow up (+/- 3 months)
  To assess blood test variables in the persistence or recurrence of LV thrombus
Quality of Life Questionnaire | From baseline to final 12 month follow up (+/- 2 months)
  Participants quality of life (QoL) will be measured using European Quality of Life-5 Dimensions - 5 levels (EQ-5D-5L) questionnaire at baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No